CLINICAL TRIAL: NCT01363908
Title: A Phase 2, Open Label, Multi-Center, Single-Dose Pharmacokinetics, and Multiple Dose Study of the Safety, Efficacy and Tolerability of SSP-004184 (SPD602) in a Pediatric Population With Transfusional Iron Overload
Brief Title: Safety, Efficacy and Pharmacokinetics of an Oral Iron Chelator Given for a Year to Pediatric Patients With Iron Overload
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to treatment stop resulting in an inability to draw conclusions from the data. Evaluation of nonclinical rat findings is ongoing.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD602-202; SSP-004184AQ (Other: Shire)
Record Dates: First submitted 2011-05-30; First posted 2011-06-02 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Transfusional Iron Overload; Beta-Thalassemia
Keywords: Beta-Thalassemia; Sickle Cell Anemia; Transfusional iron overload; Iron Overload; Iron Chelation
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell; Iron Overload

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SPD602 (26 mg/kg) (Experimental): Oral SSP-004184AQ taken once daily for 48 weeks
  Interventions: Drug: SPD602
- SPD602 (36 mg/kg) (Experimental): Oral SSP-004184AQ taken once daily for 48 weeks. Starting dose based on transfusion burden and iron overload status. Doses may range from 8-60mg/kg/day depending on clinical response.
  Interventions: Drug: SPD602
- SPD602 (16 mg/kg) (Experimental): A single dose given in the initial pharmacokinetic phase.
  Interventions: Drug: SPD602

INTERVENTIONS:
Drug: SPD602
  Other Names: SSP-004184, deferitazole

SUMMARY:
This is an open-label study to assess the pharmacokinetics, safety, efficacy and tolerability of SSP-004184AQ. The study consists of two phases: the pharmacokinetic phase, using a single 16 mg/kg dose of SSP-004184AQ; and the chronic dosing phase, during which patients will receive an additional 48 weeks of SSP-004184AQ dosing. Two age groups will be studied: 6-<12, and 12-<18 years old. The study is designed to initially assess the pharmacokinetics and safety of SSP-004184AQ in older children (adolescents, 12-<18 years old) and then if deemed safe, in younger children (6-<12 years old).

DETAILED DESCRIPTION:
Pharmacokinetic Phase: Patients will receive a single 16 mg/kg dose of SSP-004184AQ in capsule form.

Chronic Dosing Phase: Patients will receive SSP-004184AQ capsules daily for 48 weeks. Doses may range from 8-60 mg/kg/d.

ELIGIBILITY:
Inclusion Criteria

* Parents willing and able to sign the approved informed consent for their children and subjects between the ages of 6 and <18 years willing and able to provide their assent (based on institutional guidelines).
* Able to swallow whole capsules.
* Age >6 and <18 years.
* Transfusion-dependent subjects who have transfusional iron overload requiring chronic treatment with deferoxamine, deferasirox, or deferiprone. A transfusion dependent subject is defined in this study as one with a minimum transfusion history totaling more than 20 units of packed red blood cells OR a calculated iron load based on transfusion history of 200mg/kg AND a transfusion requirement of 7 or more transfusions per year; or, in subjects with sickle cell anemia, be iron overloaded but can be receiving transfusion exchange therapy in lieu of transfusions.
* In the opinion of the Investigator (and in consultation with the subject's parents), the subject is able to discontinue all existing iron chelation therapies for a minimum period of 1-5 days prior first dose of SSP-004184AQ, for the initial pharmacokinetic period of 8 days (if applicable), and for up to 49 weeks if continuing into the chronic dosing phase.
* Subjects able to have an MRI must have:

  1. liver iron concentration >2 and <30mg/g (dry weight, liver) by FerriScan® R2
  2. cardiac MRI T2* >10ms (Note: Subjects not able to have an MRI will be considered iron overloaded on the basis of serum ferritin only.)
* Serum ferritin >500ng/mL at Screening.
* Mean of the previous 3 pre-transfusion hemoglobin concentrations greater than or equal to 7.5g/dL.
* If appropriate, depending on age, female subjects of child-bearing potential need to use a medically acceptable method for birth control from screening until 30 days after the last dose of the study drug. Females of child-bearing potential must have a negative serum beta-HCG pregnancy test at the Screening Visit and a negative urine pregnancy test at the Baseline Visit. Females of child-bearing potential must agree to abstain from sexual activity that could result in pregnancy or agree to use acceptable methods of contraception.

Exclusion Criteria

* As a result of medical review, physical examination (including height and weight) or Screening investigations, the Principal Investigator considers the subject unfit for the study.
* Iron overload from causes other than transfusional hemosiderosis.
* Severe cardiac dysfunction.
* Non-elective hospitalization within the 30 days prior to Baseline testing.
* Evidence of clinically significant oral, cardiovascular, gastrointestinal, hepatic, biliary, renal, endocrine, pulmonary, neurologic, psychiatric, or skin disorder that contra-indicates dosing with SSP-004184AQ.
* Evidence of significant renal insufficiency, eg, serum creatinine above the upper limit of normal or proteinuria greater than 1 gm per day.
* Known sensitivity to any ingredient in the SSP-004184AQ formulation.
* Platelet count below 100,000/µL or absolute neutrophil count less than 1500/mm3 at Screening.
* ALT >180 IU/L at Screening.
* Use of any investigational agent within the 30 days prior to Baseline testing.
* Pregnant or lactating females.
* Cardiac left ventricular ejection fraction a) Below the locally determined normal range in the 12 months prior to screening by echocardiography or MRI or <50% at Baseline testing by MRI (echocardiograph is acceptable for LVEF if MRI information is not available).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-08-10 (Actual); Primary Completion 2014-05-13 (Actual); Study Completion 2014-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Toronto Sick Kids Hospital, Toronto, Ontario, Canada
- Italy (3):
  - Ospedale Regionale Mecrocitemie, Cagliari
  - Centro della Microcitemia e delle Anemie Congenite, Genoa
  - Thalassemia Center San Luigi Hospital, Orbassano
- Lebanon (2):
  - American University of Beirut Medical Center, Beirut
  - Chronic Care Center, Beirut
- Ege University Hospital, Izmir, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted a pharmacokinetic (PK) phase and a chronic dosing (CD) phase. A sufficient number of participants were screened to enroll 16 participants into the PK phase (8 participants per age cohort). These participants could consent to participate in the CD phase. Additional participants also participated in the CD phase.
Groups:
- 6 to <12 Year Old: During the pharmacokinetic phase, participants aged 6 to less than 12 years received a single oral dose of SPD602 16mg/kg. During the chronic dosing phase, participants commenced 48 weeks of treatment with an initial dose of SPD602 26mg/kg/day or 36mg/kg/day. Over the course of treatment, the dose could range from 8-60mg/kg/day depending on clinical response.
- 12 to <18 Year Old: During the pharmacokinetic phase, participants aged 12 to less than 18 years received a single oral dose of SPD602 16mg/kg. During the chronic dosing phase, participants commenced 48 weeks of treatment with an initial dose of SPD602 26mg/kg/day or 36mg/kg/day. Over the course of treatment, the dose could range from 8-60mg/kg/day depending on clinical response.
Period: Screening/Enrollment
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Started | 14 | 16
Completed | 13 (One participant did not receive investigational product.) | 16
Not Completed | 1 | 0
Period: Pharmacokinetic (PK) Phase
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Started | 8 (Per study design, at least 8 participants in each age cohort participated in the PK phase.) | 8 (Per study design, at least 8 participants in each age cohort participated in the PK phase.)
Completed | 8 | 8
Not Completed | 0 | 0
Period: Chronic Dosing (CD) Phase
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Started | 13 (The CD phase enrolled willing participants who completed the PK phase plus additional participants.) | 16 (The CD phase enrolled willing participants who completed the PK phase plus additional participants.)
Completed | 3 | 10
Not Completed | 10 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Patient decision | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Early study termination | 9 | 3

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set, defined as all participants who had taken at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (1.85) | 14.4 (1.78) | 11.8 (3.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of SPD602 After a Single Oral Dose
Description: The pharmacokinetic (PK) parameters of SPD602 were measured in plasma of all patients following a single capsule dose of SPD602 at 16 mg/kg at start of treatment on Day 1 and at the clinic visit on Day 2. PK blood samples were collected as follows: Pre-dose on Day 1 (within 60 minutes prior to investigational product administration) and at 0.5, 1, 2, 3, 4, 8 hours (±3 minutes) and 24 hours (±30 minutes) post-dose. Plasma concentrations of SPD602 were determined using a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. The PK parameters were determined from plasma concentration-time data for SPD602 (total) by non-compartmental analysis.
Time Frame: Day 1 and up to 24 hours post-dose
Population: The Pharmacokinetic (PK) set, defined as all participants in the Safety Analysis Set for whom the primary PK data were considered sufficient and interpretable. The Safety Analysis Set was defined as all participants who had taken at least 1 dose of investigational product. Treatment assignment was based on the treatment actually received.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 8 | 8
ng/mL | 31737.5 (10116.74) | 28300.0 (7309.88)

2. Primary Outcome: Time of Maximum Observed Plasma Concentration Sampled During a Dosing Interval (Tmax) of SPD602 After a Single Oral Dose
Description: as for outcome 1
Time Frame: Day 1 and up to 24 hours post-dose
Population: The PK set, defined as all participants in the Safety Analysis Set for whom the primary PK data were considered sufficient and interpretable.
Measure: Median (Full Range); unit: hours
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 8 | 8
hours | 1.0 [0.5 to 1.0] | 1.0 [0.6 to 2.0]

3. Primary Outcome: Area Under The Plasma Concentration-Time Curve (AUC) From The Time of Dosing to The Last Measurable Concentration (AUClast) of SPD602 After a Single Oral Dose
Description: as for outcome 1
Time Frame: Day 1 and up to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*mg/L
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 8 | 8
h*mg/L | 69.4 (27.39) | 71.6 (22.70)

4. Primary Outcome: Terminal Half-life (t1/2) of SPD602 After a Single Oral Dose
Description: as for outcome 1
Time Frame: Day 1 and up to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 8 | 8
hours | 3.7 (0.93) | 3.6 (0.97)

5. Primary Outcome: Renal Clearance (CLr) of SPD602 After a Single Oral Dose
Description: The pharmacokinetic (PK) parameters of SPD602 were measured in urine of patients following a single capsule dose of SPD602 at 16 mg/kg at start of treatment on Day 1 and at the clinic visit on Day 2. Children who could cooperate provided urine samples for PK assessment on Day 1 over 3 time intervals: 0-4, 4-8, and 8-24 hours after the last dose (continued into Day 2). Urine concentrations of SPD602 were determined using a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. The PK parameters were determined from urine concentration-time data for SPD602 (total) by non-compartmental analysis.
Time Frame: Day 1 and up to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 8 | 8
L/h | 3.6 (2.06) | 5.4 (2.38)

6. Primary Outcome: Amount Excreted Into Urine (Ue) of SPD602 After a Single Oral Dose
Description: as for outcome 5
Time Frame: Day 1 and up to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 8 | 8
mg | 227.9 (107.44) | 369.7 (140.17)

7. Primary Outcome: Fraction Of Orally Administered Drug Excreted Unchanged In Urine (fe) of SPD602 After a Single Oral Dose
Description: as for outcome 5
Time Frame: Day 1 and up to 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of total dose
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 8 | 8
percentage of total dose | 42.1 (14.34) | 52.5 (20.52)

8. Primary Outcome: Change From Baseline in Liver Iron Concentration (LIC) Assessed by FerriScan R2 Magnetic Resonance Imaging (MRI)
Description: The efficacy of SPD602 was assessed by determining LIC. Abdominal MRI data were collected by using FerriScan R2 standard procedures and used to determine LIC. A negative change from baseline indicates that LIC decreased.
Time Frame: Baseline, 24 weeks, and 48 weeks
Population: The Full Analysis Set (FAS), defined as all participants in the Safety Analysis Set who had at least 1 post-baseline primary efficacy assessment, which was considered as the LICs assessed from FerriScan R2 MRI.
Measure: Mean (Standard Deviation); unit: mg Fe/g*dw
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 10 | 15
mg Fe/g*dw
  Week 24, n=7,15 | -1.8 (2.8) | 0.8 (2.7)
  Week 48, n=2,10 | 0.8 (0.4) | -0.2 (1.8)
Statistical Analysis 1: Comparison: 6 to <12 Year Old; Analysis of 6 to <12 year olds at 24 weeks; Test type: Superiority or Other; p = 0.0781, Wilcoxon signed rank test — The P-value was from the analysis of Wilcoxon signed rank test at post-treatment time point vs baseline
Statistical Analysis 2: Comparison: 6 to <12 Year Old; Analysis of 6 to <12 year olds at 48 weeks; Test type: Superiority or Other; p = 0.5000, Wilcoxon signed rank test — The P-value was from the analysis of Wilcoxon signed rank test at post-treatment time point vs baseline
Statistical Analysis 3: Comparison: 12 to <18 Year Old; Analysis of 12 to <18 year olds at 24 weeks; Test type: Superiority or Other; p = 0.2609, Wilcoxon signed rank test — The P-value was from the analysis of Wilcoxon signed rank test at post-treatment time point vs baseline
Statistical Analysis 4: Comparison: 12 to <18 Year Old; Analysis of 12 to <18 year olds at 48 weeks; Test type: Superiority or Other; p = 0.9219, Wilcoxon signed rank test — The P-value was from the analysis of Wilcoxon signed rank test at post-treatment time point vs baseline

9. Primary Outcome: Change From Baseline in LIC Adjusted by Transfusional Iron Intake And Assessed by FerriScan R2 MRI
Description: The efficacy of SPD602 was assessed by determining LIC and adjusting for transfusional iron intake. Abdominal MRI data were collected by using FerriScan R2 standard procedures and used to determine LIC. A negative change from baseline indicates that LIC decreased.
Time Frame: Baseline, 24 weeks, and 48 weeks
Population: The FAS, defined as all participants in the Safety Analysis Set who had at least 1 post-baseline primary efficacy assessment, which was considered as the LICs assessed from FerriScan R2 MRI.
Measure: Mean (Standard Deviation); unit: mg Fe/g*dw
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 10 | 15
mg Fe/g*dw
  Week 24, n=7,15 | -8.3 (3.7) | -4.0 (3.1)
  Week 48, n=2,10 | -13.7 (5.3) | -11.9 (5.4)

10. Secondary Outcome: Change From Baseline in LIC Assessed by R2* MRI
Description: The efficacy of SPD602 was assessed by determining LIC. Abdominal MRI data were collected by using R2* standard procedures and used to determine LIC. A negative change from baseline indicates that LIC decreased.
Time Frame: Baseline, 24 weeks, and 48 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg Fe/g*dw
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 10 | 15
mg Fe/g*dw
  Week 24, n=7,15 | 0.3 (1.7) | 0.2 (1.4)
  Week 48, n=3,10 | 0.6 (4.1) | 0.3 (1.9)
Statistical Analysis 1: Comparison: 6 to <12 Year Old; Analysis of 6 to <12 year olds at 24 weeks; Test type: Superiority or Other; p = 0.6875, Wilcoxon signed-rank test — The P-value was from analysis of Wilcoxon signed-rank test at post-treatment time point vs. baseline
Statistical Analysis 2: Comparison: 6 to <12 Year Old; Analysis of 6 to <12 year olds at 48 weeks; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test — The P-value was from analysis of Wilcoxon signed-rank test at post-treatment time point vs. baseline
Statistical Analysis 3: Comparison: 12 to <18 Year Old; Analysis of 12 to <18 year olds at 24 weeks; Test type: Superiority or Other; p = 0.8181, Wilcoxon signed-rank test — The P-value was from analysis of Wilcoxon signed-rank test at post-treatment time point vs. baseline
Statistical Analysis 4: Comparison: 12 to <18 Year Old; Analysis of 12 to <18 year olds at 48 weeks; Test type: Superiority or Other; p = 0.5566, Wilcoxon signed-rank — P-value was from analysis of Wilcoxon signed-rank test at post-treatment time point vs. baseline

11. Secondary Outcome: Change From Baseline in LIC Adjusted by Transfusional Iron Intake And Assessed by R2* MRI
Description: The efficacy of SPD602 was assessed by determining LIC and adjusting for transfusional iron intake. Abdominal MRI data were collected by using R2* standard procedures and used to determine LIC. A negative change from baseline indicates that LIC decreased.
Time Frame: Baseline, 24 weeks, and 48 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg Fe/g*dw
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 10 | 15
mg Fe/g*dw
  Week 24, n=7,15 | -6.2 (2.2) | -4.6 (3.4)
  Week 48, n=3,10 | -9.1 (5.6) | -11.4 (5.2)

12. Secondary Outcome: Change From Baseline in Cardiac Iron Load Assessed by T2* MRI
Description: The efficacy of SPD602 was assessed by determining cardiac iron load. Cardiac MRI data were collected by using T2* standard procedures and used to determine iron load. A negative change from baseline indicates that iron load increased.
Time Frame: Baseline, 24 weeks, and 48 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 10 | 15
milliseconds
  Week 24, n=7,15 | -9.63 (10.766) | -6.27 (13.731)
  Week 48, n=3,10 | -10.60 (20.893) | -9.40 (14.693)
Statistical Analysis 1: Comparison: 6 to <12 Year Old; Analysis of 6 to <12 year olds at 24 weeks; Test type: Superiority or Other; p = 0.0475, paired t test — The P-value was from paired t test for log-transformed data at post-treatment time point vs. baseline
Statistical Analysis 2: Comparison: 6 to <12 Year Old; Analysis of 6 to <12 year olds at 48 weeks; Test type: Superiority or Other; p = 0.4410, paired t test — The P-value was from paired t test for log-transformed data at post-treatment time point vs. baseline; The P-value was from paired t test for log-transformed data at post-treatment time point vs. baseline
Statistical Analysis 3: Comparison: 12 to <18 Year Old; Analysis of 12 to <18 year olds at 24 weeks; Test type: Superiority or Other; p = 0.0417, paired t test — The P-value was from paired t test for log-transformed data at post-treatment time point vs. baseline
Statistical Analysis 4: Comparison: 12 to <18 Year Old; Analysis of 12 to <18 year olds at 48 weeks; Test type: Superiority or Other; p = 0.0409, paired t test — The P-value was from paired t test for log-transformed data at post-treatment time point vs. baseline

13. Secondary Outcome: Change From Baseline in Serum Ferritin
Description: Serum ferritin levels were assessed to determine if a participant was a successful responder and were determined from serum biochemistry analyses conducted at the central laboratories. A negative change from baseline indicates that serum ferritin decreased.
Time Frame: Baseline, 24 weeks, and 48 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Number analyzed (Participants) | 10 | 15
ng/mL
  Week 24, n=7,15 | 73.19 (706.423) | -981.49 (1694.314)
  Week 48, n=3,10 | -590.21 (843.249) | -1119.90 (1503.732)
Statistical Analysis 1: Comparison: 6 to <12 Year Old; Analysis of 6 to <12 year olds at 24 weeks; Test type: Superiority or Other; p = 0.9901, paired t test — The P-value was from paired t test for log-transformed data at post-treatment time point vs. baseline
Statistical Analysis 2: Comparison: 6 to <12 Year Old; Analysis of 6 to <12 year olds at 48 weeks; Test type: Superiority or Other; p = 0.3039, paired t test — The P-value was from paired t test for log-transformed data at post-treatment time point vs. baseline
Statistical Analysis 3: Comparison: 12 to <18 Year Old; Analysis of 12 to <18 year olds at 24 weeks; Test type: Superiority or Other; p = 0.0044, paired t test — The P-value was from paired t test for log-transformed data at post-treatment time point vs. baseline
Statistical Analysis 4: Comparison: 12 to <18 Year Old; Analysis of 12 to <18 year olds at 48 weeks; Test type: Superiority or Other; p = 0.0395, paired t test — The P-value was from paired t test for log-transformed data at post-treatment time point vs. baseline

ADVERSE EVENTS:
Arm/Group | 6 to <12 Year Old | 12 to <18 Year Old
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 13/13 | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 to <12 Year Old (N=13) | 12 to <18 Year Old (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (5)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 3 (7)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (7)
Vomiting (Gastrointestinal disorders) | 4 (6) | 5 (5)
Asthenia (General disorders) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (2) | 2 (3)
Pyrexia (General disorders) | 2 (2) | 5 (8)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (2)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (5)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Glucose tolerance test abnormal (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (3)
Spleen palpable (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (10) | 8 (13)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Hyporeflexia (Nervous system disorders) | 0 (0) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 2 (3)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (3) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hyperaemia (Vascular disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early because of non-clinical safety results. As such, not all subjects completed the study. The available efficacy data were summarized and analyzed as specified in the SAP; however, no efficacy conclusions could be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.